CLINICAL TRIAL: NCT04095351
Title: Connective Tissue Diseases and Lung Manifestations Prospective Trial With Focus on Systemic Sclerosis (Colipris)
Brief Title: Connective Tissue Diseases and Lung Manifestations
Acronym: Colipris
Status: Recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 20190506-2003
Record Dates: First submitted 2019-09-13; First posted 2019-09-19 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2019-09

CONDITIONS: Connective Tissue Diseases; Interstitial Lung Disease; Systemic Sclerosis
MeSH Terms: conditions — Connective Tissue Diseases; Lung Diseases, Interstitial; Scleroderma, Systemic | interventions — Respiratory Function Tests; Diagnostic Imaging; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — From each patient with proven systemic sclerosis one serum vial of 10 ml and 2 EDTA vials à 10 ml will be taken. Peripheral blood mononuclear cells are isolated from the EDTA blood samples, an stored at -80°C.The serum samples will be centrifuged and the resulting serum is collected in cryovials and stored at -80 °C until measurement. Samples and data will be stored and archived central according to the new standards of the biobank facility of the medical university of Innsbruck.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Pulmonary function test — Spirometry or plethysmography, measurement of diffusion capacity
Diagnostic Test: Imaging — Thoracic ultrasound, HRCT as scheduled within routine clinical examinations, echocardiography
Biological: Blood sampling — Standard laboratory test for CTDs as part of routine clinical examination

SUMMARY:
Despite a number of prospective studies already initiated in the past years, the current epidemiology and course of interstitial lung disease (ILD) and pulmonary hypertension (PH) in patients with connective tissue disease (CTD) is still not well defined, particularly regarding its prevalence, incidence and the management of a broad spectrum of disease presentations.

Major challenges include the identification of patients with progressive disease, the appropriate time point of therapeutic intervention and the underlying driver of disease (inflammatory or pro-fibrotic stimulus or both?).

To address these issues in Western Austria, a progressive registry of patients with CTD exploring routine clinical and pathophysiological characteristics of ILD and PH will be conducted. This multidisciplinary, prospective and observational registry aims to collect comprehensive clinical data on incidence, prevalence and course of disease regarding all PH and ILD presentations in a real-world setting.

DETAILED DESCRIPTION:
Specifically, this registry will collect demographic data, disease-related clinical data, routine laboratory values (including antibody-profile and iron status), diagnostic procedures, significant comorbidities, therapeutic managements (e.g. thoracic ultrasound, HRCT), and disease outcomes over 10 years.

In addition, blood biobank samples for translational research will be collected in a subgroup of patients with systemic sclerosis over serial time points to study the systemic inflammatory and profibrotic phenotype of patients. In summary, this registry will monitor the disease course of pulmonary manifestations of patients with CTD and may be hypothesis-generating and provide new insights in underlying inflammatory/pro-fibrotic patterns.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are adult patients (≥18 years) diagnosed with CTD with signed informed consent.

Exclusion Criteria:

* Exclusion criteria are patients with a serious co-morbidity interfering with the course of interstitial lung disease or pulmonary hypertension.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real-life cohort of CTD patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2034-10-01 (Estimated)

PRIMARY OUTCOMES:
Decline in forced vital capacity | 1 year
  Absolute decline from baseline in forced vital capacity percent predicted. Lung function tests are performed by a trained professional.
Increase in the modified Rodnan Skin Score | 1 year
  Change in the modified Rodnan Skin Score from baseline of >5 Points assessed by a trained professional
Decline in Diffusion capacity for carbon monoxide | 1 year
  Absolute decline from baseline in diffusion capacity for carbon monoxide in percent measured. Lung function tests are performed by a trained professional.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Löffler-Ragg, Prof. MD, Principal Investigator — Medical University Innsbruck, Department Internal Medicine
Locations (1):
- Medical University Innsbruck, Department of Internal Medicine II, Innsbruck, Austria